CLINICAL TRIAL: NCT00084942
Title: A Phase II Study of Gemcitabine in Combination With Capecitabine in Advanced Cholangiocarcinoma
Brief Title: Gemcitabine and Capecitabine in Treating Patients With Advanced and/or Inoperable Cholangiocarcinoma or Carcinoma of the Gallbladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Miland Javle, MD, Roswell Park Cancer Institute
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000367107; RPCI-RPC-0205
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer
Keywords: cholangiocarcinoma of the gallbladder; recurrent gallbladder cancer; unresectable gallbladder cancer; cholangiocarcinoma of the extrahepatic bile duct; recurrent extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine with capecitabine in treating patients who have advanced and/or inoperable cholangiocarcinoma or carcinoma (cancer) of the gallbladder.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with advanced and/or inoperable cholangiocarcinoma or carcinoma of the gallbladder treated with gemcitabine and capecitabine.

Secondary

* Determine time to disease progression and overall survival of patients treated with this regimen.
* Determine quality of life of patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and at weeks 3, 6, 9, and 12.

Patients are followed monthly.

PROJECTED ACCRUAL: A total of 9-17 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed cholangiocarcinoma or carcinoma of the gallbladder

  * Advanced and/or inoperable disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 2 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin < 3 mg/dL

Renal

* Creatinine ≤ 1.6 mg/dL

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to study drugs
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 weeks since prior chemotherapy and recovered
* No more than 1 prior chemoembolization OR chemoradiotherapy regimen for locally advanced biliary tract cancer
* No other prior chemotherapy (except adjuvant therapy)

Endocrine therapy

* Not specified

Radiotherapy

* See Chemotherapy
* More than 4 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Primary Completion 2004-05 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, MD, Principal Investigator — Roswell Park Cancer Institute; John Gibbs, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States